CLINICAL TRIAL: NCT00253682
Title: Cardiac Status of HAART Exposed Infants of HIV-Infected Mothers (CHAART I)
Brief Title: Effects of Highly Active Anti-Retroviral Therapy on Cardiovascular Health in Infants of HIV-Infected Mothers
Acronym: CHAART-1
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Baylor College of Medicine (Other); University of Illinois at Chicago (Other); Clinical Trials & Surveys Corp (C-TASC) (Industry); Columbia University (Other); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Steven E. Lipshultz, MD, Voluntary Professor, University of Miami
Other Study IDs: 342; R01HL072705 (NIH)
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; HIV Infections; Cardiomyopathy, Hypertrophic
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; HIV Infections; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples were collected for analysis of cardiac biomarkers high sensitivity C REactive PRotein (hsCRP) and N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: HIV-uninfected infants born to HIV-infected women with in-utero exposure to HIghly Active Ani-Retroviral Therapy (HAART) who were enrolled in the Women and Infants Transmission Study (WITS).
- 2: Historical cohort of HIV-uninfected infants born to HIV-infected women from the Pediatric Pulmonary and Cardiovascular Complications of HIV Study (P2C2 HIV) who were not exposed to HAART.

SUMMARY:
This study will determine the impact of highly active antiretroviral therapy (HAART) on the developing cardiovascular system, the evolution of HAART-associated cardiovascular changes over time, and the association between cardiovascular measurements with HAART exposure.

DETAILED DESCRIPTION:
BACKGROUND:

HIV-infected pregnant women frequently receive HAART, which is associated with reduced maternal-fetal transmission of HIV infection. This has resulted in a rapidly increasing number of seroreverters (HIV-uninfected infants born to HIV-infected women), representing the majority of infants in the United States exposed to HAART. Long-term consequences and toxicities associated with this exposure are not known, but severe cardiotoxicity is suggested in animal models. This study will utilize HIV seroreverter cohorts from the NIH-sponsored Women and Infants Transmission Study (WITS) and Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infections Study (P2C2) to determine how left ventricular (LV) structure and function, serum cardiac troponin T (cTnT), serum pro brain natriuretic peptide (proBNP), and serum high sensitivity C reactive protein (hsCRP) are affected by HAART exposure. In P2C2, patients were recruited from May 1990 to January 1994 from five clinical centers in the United States.

This study was initiated in 2002 in response to a 'Request for Applications' on HAART cardiovascular toxicities.

DESIGN NARRATIVE:

This study will utilize HIV seroreverter cohorts from the NIH-sponsored WITS and P2C2 cohorts to determine how LV structure and function, cTnT, proBNP, and hsCRP are affected by HAART exposure. The p2C2 seroreverter cohort has been exposed to no antiretroviral therapy or zidovudine alone (without HAART) and has persistent significantly depressed LV contractility in comparison to normal with up to 5 years of follow-up. The WITS seroreverter cohort has been exposed mostly to HAART. This cohort will determine the incremental effect of HAART on LV structure and function by following the P2C2 protocol for assessment of LV structure and function. This study will test three hypotheses: 1) that HAART exposure results in fetal and neonatal myocardiocyte injury and death (by serial assessment of cTnT [a biomarker of acute myocardial injury] in both seroreverter cohorts); 2) that HAART exposure results in impaired myocardiocyte mitochondrial function resulting in LV dysfunction (by serial assessment of proBNP [a biomarker related to LV dysfunction], LV volume and pressure increases resulting in LV stretch, and neurohormonal activation); and 3) that HAART exposure results in accelerated atherosclerosis (by serial assessment of hsCRP [a biomarker of generalized inflammation predictive of increased subsequent coronary artery disease]). This study will determine the cardiovascular effects of HAART in seroreverters and the need for future cardiovascular follow-up and cardiovascular preventive and therapeutic trials in this rapidly expanding population.

ELIGIBILITY:
Inclusion Criteria:

* Children who are actively enrolled in the WITS study, regardless of whether or not they have been exposed to HAART therapy
* Children enrolled into this study from one of the designated WITS clinical sites
* Mothers or legal guardians understand and are willing to provide informed consent with or without the help of an interpreter

Exclusion Criteria:

* Children diagnosed with HIV infection
* Mother has maternal diabetes or phenylketonuria
* Mother has been told by a physician that she has chromosomal defects
* Mother has functional heart defects that have required medications or surgeries
* Mother received cancer chemotherapy or radiation therapy during pregnancy
* Mother used lithium carbonate, anticonvulsants, amphetamines, or angiotensin converting enzyme (ACE) inhibitors during pregnancy

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: HIV-uninfected infants born to HIV-infected women with in-utero exposure to HIghly Active Ani-Retroviral Therapy (HAART) who were enrolled in the Women and Infants Transmission Study (WITS).
  The comparison group will be a historical cohort of HIV-uninfected infants born to HIV-infected women from the Pediatric Pulmonary and Cardiovascular Complications of HIV Study (P2C2 HIV) who were not exposed to HAART.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2002-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Lipshultz, MD, Principal Investigator — University of Miami
Locations (5):
- United States (5):
  - University of Miami School of Medicine, Miami, Florida
  - University of Illinois - Chicago, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Columbia University, New York, New York
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Seeborg FO, Gay H, Schmiege LM 3rd, Bernard D, Shearer WT. Immunoglobulin G kappa [IgG kappa] and IgG lambda paraproteinemia in a child with AIDS and response to highly active antiretroviral therapy. Clin Diagn Lab Immunol. 2005 Nov;12(11):1331-3. doi: 10.1128/CDLI.12.11.1331-1333.2005. PMID 16275950
- [Background] Shearer WT. Infection versus immunity: What's the balance? J Allergy Clin Immunol. 2005 Aug;116(2):263-6. doi: 10.1016/j.jaci.2005.06.001. No abstract available. PMID 16083777
- [Background] Simbre VC, Duffy SA, Dadlani GH, Miller TL, Lipshultz SE. Cardiotoxicity of cancer chemotherapy: implications for children. Paediatr Drugs. 2005;7(3):187-202. doi: 10.2165/00148581-200507030-00005. PMID 15977964
- [Background] Lipshultz SE, Lipsitz SR, Sallan SE, Dalton VM, Mone SM, Gelber RD, Colan SD. Chronic progressive cardiac dysfunction years after doxorubicin therapy for childhood acute lymphoblastic leukemia. J Clin Oncol. 2005 Apr 20;23(12):2629-36. doi: 10.1200/JCO.2005.12.121. PMID 15837978
- [Background] Moylett EH, Hanson IC. Mechanistic actions of the risks and adverse events associated with vaccine administration. J Allergy Clin Immunol. 2004 Nov;114(5):1010-20; quiz 1021. doi: 10.1016/j.jaci.2004.09.007. PMID 15536401
- [Background] Shearer WT. Importance of technology for the future of allergy and immunology. J Allergy Clin Immunol. 2004 Aug;114(2):406-8. doi: 10.1016/j.jaci.2004.06.031. No abstract available. PMID 15316524
- [Background] Seeborg FO, Paul ME, Abramson SL, Kearney DL, Dorfman SR, Holland SM, Shearer WT. A 5-week-old HIV-1-exposed girl with failure to thrive and diffuse nodular pulmonary infiltrates. J Allergy Clin Immunol. 2004 Apr;113(4):627-34. doi: 10.1016/j.jaci.2004.01.763. PMID 15100665
- [Background] Mone SM, Gillman MW, Miller TL, Herman EH, Lipshultz SE. Effects of environmental exposures on the cardiovascular system: prenatal period through adolescence. Pediatrics. 2004 Apr;113(4 Suppl):1058-69. PMID 15060200
- [Background] Nance CL, Shearer WT. Is green tea good for HIV-1 infection? J Allergy Clin Immunol. 2003 Nov;112(5):851-3. doi: 10.1016/j.jaci.2003.08.048. No abstract available. PMID 14610469
- [Background] Al-Attar I, Orav EJ, Exil V, Vlach SA, Lipshultz SE. Predictors of cardiac morbidity and related mortality in children with acquired immunodeficiency syndrome. J Am Coll Cardiol. 2003 May 7;41(9):1598-605. doi: 10.1016/s0735-1097(03)00256-0. PMID 12742303